CLINICAL TRIAL: NCT06931223
Title: Efficacy of Gut-rain Neuromodulators in the Treatment of Functional Dyspepsia: a Randomized Controlled Study
Brief Title: Efficacy of Gut-Brain Neuromodulators for Functional Dyspepsia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shengliang Chen, Professor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RJYYXHNK-03
Record Dates: First submitted 2025-03-31; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Functioanl Dyspepsia
MeSH Terms: interventions — flupentixol, melitracen drug combination; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients were treated with Flupentixol-Melitracen (FM) plus lansoprazole for 2 weeks (Experimental)
  Interventions: Drug: Flupentixol-Melitracen + Lansoprazole
- Patients were treated with placebo plus lansoprazole for 2 weeks (Experimental)
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Flupentixol-Melitracen + Lansoprazole — Flupentixol-Melitracen and Lansoprazole for the treatment of functional dyspepsia.
  Arms: Patients were treated with Flupentixol-Melitracen (FM) plus lansoprazole for 2 weeks
Drug: Lansoprazole — Placebo and Lansoprazole for functional dyspepsia.
  Arms: Patients were treated with placebo plus lansoprazole for 2 weeks

SUMMARY:
The use of Neuromodulators is now recognized by international consensus as effective in improving Disorders of Gut-Brain Interaction (DGBIs). However, the digestive mind-body concept of therapeutic drugs is still in the experience-based treatment stage, and there is a lack of clinical studies in the field of DGBIs. Although numerous studies have been conducted to confirm the safety of Neuromodulators for the treatment of DGBIs, the current functional dyspepsia (FD) treatment is still awaiting further explorations and accumulations. In addition, neuromodulators, like Flupentixol-Melitracen (FM), are often used as a second-line treatment option for FD after the failure of acid-suppressive therapy with proton pump inhibitors, etc. However, the efficacy of conventional drugs for FD is mediocre, which often leads to recurrent and prolonged symptoms, seriously affecting patients' confidence in treatment and their quality of life, and the repeated visits to the clinic also create a huge economic burden for the society. Therefore, we conducted a clinical trial to verify whether FM can be used as the first-line therapy to improve the efficacy of FD patients.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients with primary FD who meet the diagnostic criteria for Roman IV;
2. able to complete the questionnaire, trial evaluation and sign the written informed consent.

Exclusion Criteria:

1. organic gastrointestinal diseases by gastroenteroscopy within 6 months;
2. severe insufficiency of heart, liver, kidney, lung and other important organs and with congenital diseases;
3. allergic to the drugs used in this study
4. being pregnant, lactating or planning to become pregnant;
5. are taking or have taken monoamine oxidase inhibitors within the past 5 weeks;
6. have a known risk of narrow angle glaucoma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Leuven Postprandial Distress Scale (LPDS) score | Until the end of the study, up to 14 weeks
  The LPDS questionnaire contains 8 symptoms, namely early satiation, postprandial fullness, upper abdominal bloating, epigastric pain, epigastric burning, nausea, belching, and heartburn. Each symptom was rated on a severity scale of 0-4. The mean of the early satiation, postprandial fullness, and upper abdominal bloating scores was calculated as the postprandial distress syndrome score, and the mean of the epigastric pain, epigastric burning scores was calculated as the epigastric pain syndrome. Changes in LPDS score during the treatment period were assessed.